CLINICAL TRIAL: NCT04068545
Title: Experiences With New Digital Surgical Drainage System in Thoracic Surgery
Status: Completed | Type: Observational
Sponsor: Centese, Inc. (Industry)
Collaborators: NYU Langone Health (Other)
Responsible Party: Sponsor
Other Study IDs: CRD-1675
Record Dates: First submitted 2019-08-22; First posted 2019-08-28 (Actual); Last update posted 2020-07-17 (Actual); Status verified 2020-07

CONDITIONS: Pulmonary Air Leak

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: Device: Thoraguard Surgical Drainage System — Fluid drainage following thoracic surgery

SUMMARY:
The purpose of this study is to evaluate the Thoraguard Surgical Drainage System in a real-world clinical environment. It is believed that this system will offer functional and clinical benefits over the current standard of care system for the removal of surgical fluids and air following thoracic surgery. Observations, experiences, and outcomes in a single hospital setting will be collected for the Thoraguard Surgical Drainage System.

DETAILED DESCRIPTION:
The Thoraguard System is intended for use for drainage of blood, fluids, and gases following cardiac and thoracic surgery. The system consists of an electronic control module and drainage kit (fluid collection canister and drainage line) which connect to a proprietary chest tube but may also connect to other thoracic drainage catheters. The system continuously monitors line patency, automatically clears the chest tube (when used with Thoraguard Chest Tube) and drainage line from build-up, and provides digital readings of fluid output trends. The system is battery powered with integrated suction for ease of ambulation.

Additionally, the system has patient safety alarms to notify clinical staff of unexpected events associated with postoperative drainage. These functions offer significant improvements over the current standard of care. Reliable post-operative drainage, reduced workload, and decreased variability in chest tube maintenance procedures have the potential to increase patient safety, reduce complications, and improve the patient experience.

ELIGIBILITY:
Inclusion Criteria:

* Adult (age ≥ 18)
* Patient undergoing non-emergent thoracic surgery (Sternotomy, Video-Assisted Thoracoscopic Surgery (VATS), Thoracotomy, or Robotic)
* Expected requirement for chest drain monitoring of air leak for at least 24h post-operation
* A requirement for a surgical drainage system

Exclusion Criteria:

* Emergency surgery
* Re-do surgery
* Prior thoracic surgery
* Transplant Surgery
* In the opinion of the investigator, the patient is unsuitable for the study for any other legitimate reason including incarceration, pre-existing medical or psychiatric condition, or interfering medications
* Known previous or concurrent enrollment in a clinical trial that, in the opinion of the investigator, might interfere with the objectives of this clinical trial
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Non-emergent thoracic surgery patients undergoing a procedure for one of the following: pulmonary resection, pneumectomy, or lobectomy.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2019-09-02 (Actual); Primary Completion 2020-03-30 (Actual); Study Completion 2020-05-30 (Actual)

PRIMARY OUTCOMES:
Device User Experience Survey | At study completion - approximate 6 months.
  The Device User Experience Survey is an unvalidated, Sponsor-generated questionnaire aimed to increase the Sponsor's understanding of the usability of the Thoraguard Surgical Drainage System. The questionnaire asks approximately 15 questions (includes yes/no responses, rating scales, and fill-in-the-blank sections) and is to be completed by the treating clinicians at the completion of the study. A summary of all treating clinician responses will be generated at the completion of the study to summarize the overall user experience with the device.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Zervos, MD, Principal Investigator — NYU Langone Medical Center
Locations (1):
- NYU School of Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] McGuire AL, Petrcich W, Maziak DE, Shamji FM, Sundaresan SR, Seely AJ, Gilbert S. Digital versus analogue pleural drainage phase 1: prospective evaluation of interobserver reliability in the assessment of pulmonary air leaks. Interact Cardiovasc Thorac Surg. 2015 Oct;21(4):403-7. doi: 10.1093/icvts/ivv128. Epub 2015 Jul 14. PMID 26174120
- [Background] Pompili C, Detterbeck F, Papagiannopoulos K, Sihoe A, Vachlas K, Maxfield MW, Lim HC, Brunelli A. Multicenter international randomized comparison of objective and subjective outcomes between electronic and traditional chest drainage systems. Ann Thorac Surg. 2014 Aug;98(2):490-6; discussion 496-7. doi: 10.1016/j.athoracsur.2014.03.043. Epub 2014 Jun 4. PMID 24906602
- [Background] Miller DL, Helms GA, Mayfield WR. Digital Drainage System Reduces Hospitalization After Video-Assisted Thoracoscopic Surgery Lung Resection. Ann Thorac Surg. 2016 Sep;102(3):955-961. doi: 10.1016/j.athoracsur.2016.03.089. Epub 2016 May 25. PMID 27234573